CLINICAL TRIAL: NCT05656898
Title: Comparison Between the Flapless Corticotomy Enhanced by the Later Application of Low-intensity Laser Therapy on Patient-centred Outcomes and Periodontal Health in Patients Undergoing en Masse Retraction of Upper Anterior Teeth
Brief Title: Evaluation of the Levels of Pain and Discomfort and Periodontal Status Between Two Acceleration Methods of Upper Anterior Teeth Retraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-16-2021
Record Dates: First submitted 2022-12-07; First posted 2022-12-19 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Class II Malocclusion
MeSH Terms: conditions — Overbite | interventions — Orthodontic Appliances, Fixed

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Piezosurgery pulse Low-level laser therapy (Experimental): Piezocision will be applied in this group of patients using a piezosurgery knife and after 6 weeks of initial retraction, low-level laser therapy will be applied in this group of patients using a diode laser device.
  Interventions: Device: Piezocision+GaALAs diode laser
- Piezosurgery (Experimental): Piezocision will be applied in this group of patients using a piezosurgery knife.
  Interventions: Device: Piezocision
- Traditional treatment (Active Comparator): En masse retraction in this group will be performed in a conventional method.
  Interventions: Device: Orthodontic fixed appliance

INTERVENTIONS:
Device: Piezocision+GaALAs diode laser — After seven weeks of piezosurgery, GaALAs diode laser (wavelength: 810 nm and exposure time of 10 seconds\point) 10 seconds per point will be applied on each tooth of the six maxillary anterior teeth .
  Arms: Piezosurgery pulse Low-level laser therapy
Device: Piezocision — Vertical soft-tissue incisions will be made on the buccal and palatal gingiva. One incision will be made between the roots of the six upper anterior teeth, and two incisions will be made between the upper canines and the second premolars.
  Arms: Piezosurgery
Device: Orthodontic fixed appliance — Closed nickel-titanium coil springs applying 250 g of force per side will be used for retraction of the maxillary anterior teeth.
  Arms: Traditional treatment

SUMMARY:
60 patients will be treated by extraction of maxillary first premolars by applying mini-screws between the maxillary second premolar and first molar as temporary skeletal anchorage devices (TSADs). They will be divided randomly into three groups in this trial. The prolonged duration of the treatment period can cause many side effects such as white spots, caries, periodontal diseases, and pain and discomfort. So many efforts have been made to reduce the treatment time. Many procedures have been introduced to accelerate orthodontic tooth movement, which can category as surgical or non-surgical. Piezocision is a minimally invasive surgical method for accelerating orthodontic tooth movement and shortening treatment time. Low-level laser therapy (LLLT) is one of the physical acceleration methods that have contributed to decreasing treatment time.

DETAILED DESCRIPTION:
Closed nickel-titanium coil springs applying 250 g of force per side will be used for retraction of the maxillary anterior teeth.

The en-masse retraction will be obtained with two nickel-titanium coil springs placed between the mini-implants and the soldered hooks in a direction approximately parallel to the occlusal plane, a force of 250 g will be applied on each side to perform en-masse retraction. The retraction will be stopped when a Class I canine relation is achieved and a good incisor relation is obtained or spaces lateral to canines are closed.

Regarding the Piezocision, vertical soft-tissue incisions will be made on the buccal and palatal gingiva. One incision will be made between the roots of the six upper anterior teeth, and two incisions will be made between the upper canines and the second premolars. The incisions will be 5 mm long and start 4 mm apical to the interdental papilla. Then a piezosurgery knife will be inserted to perform the cortical alveolar incisions with 3-mm in-depth and 8 mm in length. No suturing will be needed.

Regarding the piezocision with the later application of low-level laser therapy (LLLT):

After seven weeks of piezosurgery, GaALAs diode laser (wavelength: 810 nm and exposure time of 10 seconds\point) 10 seconds per point will be applied on each tooth of the six maxillary anterior teeth according to this protocol: the root will be divided theoretically into 2 halves; gingival and cervical, and the laser will be applied in the centre of each half from both buccal and palatal sides which means 4 application points and total energy of 16 Joules per tooth. The LLLT will be applied 5 times in the first month of en masse retraction. After that, the irradiation will be repeated every two weeks, until the class, I canine relationship will be achieved and/or spaces lateral to incisors were closed

ELIGIBILITY:
Inclusion Criteria:

1. Adult healthy patients, Male and female, Age range: 17-28 years.
2. Class II Division 1 malocclusion :

   * Mild/moderate skeletal Class II (sagittal discrepancy angle ≤7)
   * Overjet ≤10
   * Normal or excessive facial height (Clinically and then cephalometrically assessed using these three angles: mandibular/cranial base angle, maxillary/mandibular plane angle, and facial axis angle)
   * Mild to moderate crowding ≤ 4
3. Permanent occlusion.
4. Existence of all the upper teeth (except third molars).
5. Good oral and periodontal health:

   * Probing depth < 4 mm
   * No radiographic evidence of bone loss.
   * Gingival index ≤ 1
   * Plaque index ≤ 1

Exclusion Criteria:

1. Medical problems that affect tooth movement (corticosteroid, nonsteroidal anti-inflammatory drugs (NSAIDs), …)
2. Presence of primary teeth in the maxillary arch
3. Missing permanent maxillary teeth (except third molars).
4. Poor oral hygiene or Current periodontal disease:

   * Probing depth ≥ 4 mm
   * radiographic evidence of bone loss
   * Gingival index > 1
   * Plaque index > 1
5. The patient had previous orthodontic treatment

Ages: 17 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Change in the levels of pain during the first month of treatment assessed by the VAS | Time 1: 12 hours, Time 2: Day 1, Time 3: Day 3, Time 4: Day 7, Time 5: Day 14, following the commencement of the retraction.
  Assessment will be performed using questionnaires via the Visual Analog scale (VAS). The Visual Analog Scale is a 100 mm horizontal line with two focal points at its beginning and end (0: no pain - 100: the worst pain).
Change in the levels of pain during the third month of treatment assessed by the VAS | Time 1: 12 hours, Time 2: Day 1, Time 3: Day 3, Time 4: Day 7, Time 5: Day 14, following the commencement of the retraction.
  Assessment will be performed using questionnaires via the Visual Analog Scale (VAS). The Visual Analog Scale is a 100 mm horizontal line with two focal points at its beginning and end (0: no pain - 100: the worst pain).
Change in the levels of discomfort during the first month of treatment assessed by the VAS | Time 1: 12 hours, Time 2: Day 1, Time 3: Day 3, Time 4: Day 7, Time 5: Day 14, following the commencement of the retraction.
  Assessment will be performed using questionnaires via the Visual Analog scale (VAS). The Visual Analog Scale is a 100 mm horizontal line with two focal points at its beginning and end (0: no pain - 100: the worst pain).
Change in the levels of discomfort during the third month of treatment assessed by the VAS | Time 1: 12 hours, Time 2: Day 1, Time 3: Day 3, Time 4: Day 7, Time 5: Day 14, following the commencement of the retraction.
  Assessment will be performed using questionnaires via the Visual Analog scale (VAS). The Visual Analog Scale is a 100 mm horizontal line with two focal points at its beginning and end (0: no pain - 100: the worst pain).
Change in the levels of swelling during the first month of treatment assessed by the VAS | Time 1: 12 hours, Time 2: Day 1, Time 3: Day 3, Time 4: Day 7, Time 5: Day 14, following the commencement of the retraction.
  Assessment will be performed using questionnaires via the Visual Analog scale (VAS). The Visual Analog Scale is a 100 mm horizontal line with two focal points at its beginning and end (0: no pain - 100: the worst pain).
Change in the levels of swelling during the third month of treatment assessed by the VAS | Time 1: 12 hours, Time 2: Day 1, Time 3: Day 3, Time 4: Day 7, Time 5: Day 14, following the commencement of the retraction.
  Assessment will be performed using questionnaires via the Visual Analog scale (VAS). The Visual Analog Scale is a 100 mm horizontal line with two focal points at its beginning and end (0: no pain - 100: the worst pain).
Change in the levels of eating difficulty during the first month of treatment assessed by the VAS | Time 1: 12 hours, Time 2: Day 1, Time 3: Day 3, Time 4: Day 7, Time 5: Day 14, following the commencement of the retraction.
  Assessment will be performed using questionnaires via the Visual Analog scale (VAS). The Visual Analog Scale is a 100 mm horizontal line with two focal points at its beginning and end (0: no pain - 100: the worst pain).
Change in the levels of eating difficulty during the third month of treatment assessed by the VAS | Time 1: 12 hours, Time 2: Day 1, Time 3: Day 3, Time 4: Day 7, Time 5: Day 14, following the commencement of the retraction.
  Assessment will be performed using questionnaires via the Visual Analog scale (VAS). The Visual Analog Scale is a 100 mm horizontal line with two focal points at its beginning and end (0: no pain - 100: the worst pain).
Change in the levels of satisfaction assessed by the VAS | These levels will be assessed only at day 14 of month 3 following the commencement of the retraction.
  Assessment will be performed using questionnaires via the Visual Analog scale (VAS). The Visual Analog Scale is a 100 mm horizontal line with two focal points at its beginning and end (0: no pain - 100: the worst pain).
Recommendation of the procedure to a friend | This question is going to be posed only at day 14 of month 3 following the commencement of the retraction.
  Patients are asked if they would recommend the procedure to a friend. This question is going to be answered by "Yes" or "No", i.e., dichotomous scale.

CONTACTS AND LOCATIONS:
Overall Officials: Mudar Mohammad Mousa, DDS, Principal Investigator — Department of orthodontics, Damascus University, Syria; Mohammad Y. Hajeer, DDS,MSc,PhD, Study Director — Department of orthodontics, Damascus University, Syria
Locations (1):
- University of Damascus, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alfawal AMH, Hajeer MY, Ajaj MA, Hamadah O, Brad B, Latifeh Y. Evaluation of patient-centered outcomes associated with the acceleration of canine retraction by using minimally invasive surgical procedures: A randomized clinical controlled trial. Dent Med Probl. 2020 Jul-Sep;57(3):285-293. doi: 10.17219/dmp/120181. PMID 32909702
- [Background] Mousa MM, Hajeer MY, Burhan AS, Almahdi WH. Evaluation of patient-reported outcome measures (PROMs) during surgically-assisted acceleration of orthodontic treatment: a systematic review and meta-analysis. Eur J Orthod. 2022 Dec 1;44(6):622-635. doi: 10.1093/ejo/cjac038. PMID 35796046
- [Background] Charavet C, Lecloux G, Bruwier A, Rompen E, Maes N, Limme M, Lambert F. Localized Piezoelectric Alveolar Decortication for Orthodontic Treatment in Adults: A Randomized Controlled Trial. J Dent Res. 2016 Aug;95(9):1003-9. doi: 10.1177/0022034516645066. Epub 2016 Apr 29. PMID 27129491
- [Background] Lombardo L, Ortan YO, Gorgun O, Panza C, Scuzzo G, Siciliani G. Changes in the oral environment after placement of lingual and labial orthodontic appliances. Prog Orthod. 2013 Sep 11;14:28. doi: 10.1186/2196-1042-14-28. PMID 24326120
- [Background] Gibreal O, Hajeer MY, Brad B. Evaluation of the levels of pain and discomfort of piezocision-assisted flapless corticotomy when treating severely crowded lower anterior teeth: a single-center, randomized controlled clinical trial. BMC Oral Health. 2019 Apr 16;19(1):57. doi: 10.1186/s12903-019-0758-9. PMID 30991984